CLINICAL TRIAL: NCT06774482
Title: Evaluation of Toxicity and Outcomes of Different Therapeutic Strategies in Patients With Uterine Neoplasms Treated With Radiotherapy at the Sant'Orsola Polyclinic in Bologna.
Brief Title: Evaluation of Toxicity and Outcomes of Different Therapeutic Strategies in Patients With Uterine Neoplasms
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ESTHER
Record Dates: First submitted 2024-12-01; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: Uterine Neoplasms
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The single-center observational study aims to collect data related to the radiation treatment of uterine neoplasms. The purpose of the study is to systematically gather data on radiation treatment in uterine neoplasms in order to evaluate tumor response and potential toxicity in relation to dosages, fractionation, and techniques used, as well as the combination with other therapies and the characteristics of the disease.

Additionally, collecting data on both the characteristics of the disease and patients' comorbidities in a large sample may allow for the evaluation of any possible correlation with radiation-induced toxicities, with the aim of being able to predict and prevent them in a personalized manner in the future.

Therefore, the study's goal is to evaluate tumor response and any potential toxicity after radiotherapy treatment in relation to treatment settings, dosages, and techniques used, both for new diagnoses and for cases already diagnosed and treated from 01/01/2000 onwards at the Radiotherapy Unit of Sant'Orsola-Malpighi Polyclinic.

The structured collection of data necessary for the evaluation of the objectives will cover the observation period from 01/01/2000 to 15/12/2030, for a total of approximately 5000 patients.

DETAILED DESCRIPTION:
Uterine neoplasms include endometrial cancer and cervical cancer. The former is the fourth most common cancer in women in Europe, while cervical cancer is the second most common cancer worldwide, especially in countries where population screening is not available.

Therapy for both is, in most cases, multimodal; the main therapeutic options include surgery, systemic therapy, and radiotherapy. The various treatments may play a role as primary, adjuvant, or neoadjuvant therapy depending on the neoplasm being treated and the strategy adopted in each case.

Regarding radiotherapy, it can be used alone or more frequently in combination with other treatments, especially in the radical treatment of cervical cancer. Radiotherapy may also play a role in metastatic disease, both with curative intent and to alleviate symptoms.

Dosages, fractionation, and techniques vary depending on the type of neoplasm being treated and the purpose of the therapy (adjuvant, neoadjuvant, radical, or palliative), as do the potential acute and late toxicities in relation to the characteristics of the treatment.

The aim of the study is to systematically collect data related to radiation treatment in uterine neoplasms to evaluate outcomes in relation to dosages, fractionation, and techniques used, the combination with other therapies, and the characteristics of the disease.

Moreover, collecting data on both the disease characteristics and treatments in a large sample may make it possible to evaluate any possible correlation with radiation-induced toxicities, in order to predict and prevent them in a personalized way in the future.

Patients enrolled in all phases of the study will not experience any direct benefit or harm from it, as it is solely a data collection effort. On the contrary, this data could lead to new knowledge that may improve the future management of the analyzed neoplastic diseases.

Thus, the goal of the study is to evaluate outcomes after radiotherapy treatment in relation to treatment settings, dosages, and techniques used, both for newly diagnosed cases and for those already diagnosed and treated since 01/01/2000 at the Radiotherapy Unit of the Sant'Orsola Polyclinic.

The structured collection of data necessary to evaluate the objectives will cover the observation period from 01/01/2000 to 15/12/2030, involving approximately 5000 patients (3000 for the retrospective phase and 2000 for the prospective phase).

The study is observational, retrospective and prospective, single-center, and spontaneous.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged ≥ 18 years, with a new or previous diagnosis of malignant uterine neoplasm, starting from 01/01/2000, treated at the Radiotherapy Unit of the Sant'Orsola Polyclinic
* Obtaining informed consent

Exclusion Criteria:

* Patients with a new or previous diagnosis of malignant uterine neoplasm who choose not to undergo radiation treatment at the Radiotherapy Unit of the Sant'Orsola Polyclinic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients, aged ≥ 18 years, with a new or previous diagnosis of malignant uterine neoplasm
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Local disease recurrence | From the end of therapy to the last follow-up at 12 months
  To evaluate the outcome, particularly in terms of local disease recurrence, after radiation treatment of uterine neoplasms, in relation to the treatment setting, dosages, and techniques used, both for newly diagnosed neoplasms and for cases already diagnosed and treated since 01/01/2000 at the Sant'Orsola Polyclinic, Bologna University Hospital.

SECONDARY OUTCOMES:
Acute toxicity | immediate to 6 months after radiotherapy
  acute toxicity after radiotherapy, evaluated according to CTCAE v.5
Late toxicity | from 6 months after radiotherapy, through study completion, an average of 1 year
  late toxicity after completion of treatments, evaluated according to CTCAE v.5
Incidence of retreatments and their characteristics | During follow ups through study completion, an average of 1 year
Disease-free survival of the patients | During the follow-ups, up to the last one at 12 months
  Disease-free survival assessed based on the presence or absence of local, nodal, or metastatic recurrences
Overall survival | From enrollment to the last follow-up ar 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Giuseppe Morganti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy